CLINICAL TRIAL: NCT01837485
Title: Evaluation of the Effects of Lactol Probiotic in Comparison With Placebo on Symptoms of Irritable Bowel Syndrome
Brief Title: Probiotics in the Treatment of Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Najafabad Branch (Other)
Responsible Party: Principal Investigator, Mozhdeh Zahiri, Dr., Islamic Azad University, Najafabad Branch
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15010101882058
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Functional gastrointestinal disorders; Gut flora; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactol (Experimental)
  Interventions: Drug: Lactol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactol — The Symbiotic Lactol® (Bioplus Life Sciences Pvt.) was applied 3 times a day for 3 months. Lactol is composed of the followings; Lactobacillus Sporogenes (15 × 107 Spores), Fructo-Oligosaccharides, Microcrystalline Cellulose, Sodium starch Glycolate, Povidone, Hypermellose Stearate, Sillicon Dioxide, and Propylene Glycol.
  Arms: Lactol
Drug: Placebo — Placebo pill was applied 3 times a day for 3 months
  Arms: Placebo

SUMMARY:
Some evidences have shown that probiotics are effective in the treatment of irritable bowel syndrome. Because few evidences are available in our population, we investigated if probiotics are effective in our patients as well. We hypothesize that the probiotic Lactol which contains Lactobacillus Sporogenes reduces the symptoms of irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* diagnosis of IBS based on the Rome III criteria
* willingness to participate

Exclusion Criteria:

* receiving other probiotics compound during the study
* receiving antibiotics during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | Up to 3 months
  Abdominal pain was assessed by Rome III questionnaire at baseline and then after 3 months.
Constipation | Up to 3 months
  Constipation was assessed by Rome III questionnaire at baseline and then after 3 months.
Diarrhea | Up to 3 months
  Diarrhea was assessed by Rome III questionnaire at baseline and then after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mozhdeh Zahiri, MD, Principal Investigator — Islamic Azad University, Najafabad Branch
Locations (1):
- Shariati Hospital, Isfahan, Isfahan, Iran